CLINICAL TRIAL: NCT05838014
Title: The Effect of Sleep Deprivation on Whole-body Heat Loss in Young and Older Men During Exercise in Hot, Dry Conditions
Brief Title: Acute Sleep Deprivation on Whole-body Heat Exchange During Exercise-heat Stress in Young and Older Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Professor, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HEPRU-2023-01
Record Dates: First submitted 2023-03-30; First posted 2023-05-01 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Thermoregulation; Sleep Disturbance; Heat Exchange; Aging; Exercise
Keywords: Heat stress; Sleep; Aging; Heat dissipation; Physical activity
MeSH Terms: conditions — Parasomnias; Motor Activity; Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: Each participant will complete two exercise trials in a hot, dry environment (40°C, 15% relative humidity) where they will perform three 30 min bouts of exercise at incrementally increasing metabolic heat loads (each separated by a 15-min rest) following a period of either (i) normal sleep or (ii) 24 h of sleep deprivation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal sleep (Active Comparator): Participants will complete three 30-minute bouts of semi-recumbent cycling at incrementally increasing fixed metabolic heat loads (150, 200 and 250 W/m2) in a hot, dry condition (40°C, 15% relative humidity). Each exercise bout will be separated by a 15 minute period of rest, with the final recovery 1 hour in duration. Exercise will commence between the hours of 7 AM and 9 AM following a period of normal sleep (~8 hours) (Control condition).
  Interventions: Other: Normal sleep
- Sleep deprivation (Experimental): Participants will complete three 30-minute bouts of semi-recumbent cycling at incrementally increasing fixed metabolic heat loads (150, 200 and 250 W/m2) in a hot, dry condition (40°C, 15% relative humidity). Each exercise bout will be separated by a 15 minute period of rest, with the final recovery 1 hour in duration. Exercise will commence between the hours of 7 AM and 9 AM following a period of 24 hour of sleep deprivation (Sleep deprivation condition).
  Interventions: Other: Sleep deprivation

INTERVENTIONS:
Other: Sleep deprivation — Participants will undertake a period of 24 hours of total sleep deprivation prior to completing exercise
  Arms: Sleep deprivation
Other: Normal sleep — Participants will undertake ~8 hours of normal sleep prior to completing exercise
  Arms: Normal sleep

SUMMARY:
Sleep deprivation has long been thought to modulate thermoregulatory function. Seminal work on sleep deprivation and thermoregulation has demonstrated that sleep-deprived individuals experience greater elevations in core temperature during exercise-heat stress due to reductions in the activation of local heat loss responses of cutaneous vasodilation and sweating. However, it remains unclear 1) if reductions in local heat loss responses would compromise whole-body heat loss (evaporative + dry heat exchange) and 2) if differences exist, are they dependent on the heat load generated by exercise (increases in metabolic rate augments the rate that heat must be dissipated by the body). Further, much of the understanding of the effects of sleep deprivation on thermoregulation has been limited to assessments in young adults. Studies show that aging is associated with reduction in cutaneous vasodilation and sweating that compromise whole-body heat loss exacerbating body heat storage during moderate- and especially more vigorous-intensity exercise in the heat. However, it remains unclear if sleep deprivation may worsen this response in older adults.

The purpose of this study is therefore to evaluate the effects of sleep-deprivation on whole-body total heat loss during light, moderate, and vigorous exercise-heat stress and to assess if aging may mediate this response. To achieve this objective, direct calorimetry will be employed to measure whole-body total heat loss in young (18-30 years) and older (50-65 years) men during exercise at increasing, fixed rates of metabolic heat production of 150 (light), 200 (moderate), and 250 W/m2 (vigorous) in dry heat (40°C, ~15% relative humidity) with and without 24 hours of sleep deprivation.

ELIGIBILITY:
Inclusion Criteria:

* healthy young (18-30 years) and older males (50-65 years)
* non-smoking
* English or French speaking
* ability to provide informed consent

Exclusion Criteria:

* presence of chronic diseases (e.g., hypertension, diabetes)
* acute illness (e.g., flu, COVID-19)
* physical restriction limiting physical activity (e.g., severe arthritis, etc.)
* use of medication judged by the patient or investigators to make participation in this study inadvisable
* engaged in regular endurance training

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Evaporative heat loss | End of each exercise bout (average of last 5 minutes)
  Evaporative heat loss as assessed using a direct air calorimeter
Whole-body heat loss | End of each exercise bout (average of last 5 minutes)
  Net heat loss (dry plus/minus evaporative heat exchange) as assessed using a direct air calorimeter

SECONDARY OUTCOMES:
Dry heat loss | End of each exercise bout (average of last 5 minutes)
  Total dry heat loss as assessed using a direct air calorimeter
Body heat storage | Each 30 minute exercise bout and sum of all three exercise bouts
  Change in body heat storage (i.e., amount of heat stored in the body) calculated as the temporal summation of metabolic heat production and net heat loss
Core temperature | End of each exercise bout (average of last 5 minutes)
  Rectal temperature measured as an index of core temperature
Change in core temperature | End of each exercise bout (average of last 5 minutes)
  Change in rectal temperature from baseline resting
Heart rate | End of each exercise bout (average of last 5 minutes)
  Measured continuously using a heart rate monitor
Heart rate reserve | End of each exercise bout (average of last 5 minutes)
  Percentage of the difference between the peak heart rate
Local sweat rate (forearm, scapula) | End of each exercise bout (average of last 5 minutes)
  Sweat production assessed using ventilated capsule technique
Skin temperature | End of each exercise bout (average of last 5 minutes)
  Skin temperature measured continuously at 4-sites (chest, upper arm, thigh, calf) with mean value calculated as weighted value of 4 sites - bicep, 30%; chest, 30%; thigh, 20%; and calf, 20%.
Skin temperature (change) | End of each exercise bout (average of last 5 minutes)
  Change in skin temperature from baseline resting as assessed at 4-sites (chest, upper arm, thigh, calf) with mean value calculated as weighted value of 4 sites - bicep, 30%; chest, 30%; thigh, 20%; and calf, 20%.
Thermal comfort scale | End of the 30 minute resting baseline period, end of each 30 minute exercise bout, end of each 15 minute rest period, and 1 hour after final exercise period.
  Thermal comfort assessed via a self-report questionnaire upon verbal prompting (4-point scale; 1: comfortable to 4: very uncomfortable)
Thermal sensation | End of the 30 minute resting baseline period, end of each 30 minute exercise bout, end of each 15 minute rest period, and 1 hour after final exercise period.
  Thermal sensation assessed via a self-report questionnaire upon verbal prompting (7-point scale; 0: neutral to 7: extremely hot)
Thirst sensation | End of the 30 minute resting baseline period, end of each 30 minute exercise bout, end of each 15 minute rest period, and 1 hour after final exercise period.
  Thirst sensation assessed via a self-report questionnaire upon verbal prompting (9-point scale; 1: not thirsty at all to 9: very, very thirsty)
Rating of perceived exertion | End of the 30 minute resting baseline period, end of each 30 minute exercise bout, end of each 15 minute rest period, and 1 hour after final exercise period.
  Perceived exertion assessed via a self-report questionnaire upon verbal prompting (6: no exertion at all to 20: maximal exertion)
Stanford sleep scale | End of the 30 minute resting baseline period, end of each 30 minute exercise bout, end of each 15 minute rest period, and 1 hour after final exercise period.
  Symptoms of tiredness assess via a self-report questionnaire upon verbal prompting (How sleepy are you?) ranging from "feeling active, vital, alert, or wide awake" to "no longer fighting sleep, sleep onset soon, having dream-like thoughts"
Variables of heart rate variability | End of each exercise (average of last 5 minutes)
  Measures of variability computed from the time, frequency, time-frequency, scale-invariant, entropy, and other nonlinear domains (R-R interval data extracted from the electrocardiogram)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available with approved analysis plan and signed access agreement
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Following publication of the main study (report(s)
Access Criteria: Approved analysis plan and signed access agreement

REFERENCES:
- [Derived] Koetje NJ, Kirby NV, O'Connor FK, Richards BJ, Janetos KT, Ioannou LG, Kenny GP. Effect of 24-h Sleep Deprivation on Whole-Body Heat Loss in Older Males during Exercise in the Heat. Med Sci Sports Exerc. 2025 Dec 1;57(12):2715-2723. doi: 10.1249/MSS.0000000000003812. Epub 2025 Jul 7. PMID 40623158